CLINICAL TRIAL: NCT05649397
Title: Effects of Cervical Spine Manipulation on Proprioception, Blood Pressure and Respiratory Rate in Patients With Mechanical Neck Pain
Brief Title: Effects of Cervical Spine Manipulation in Patients With Mechanical Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC- 01395 Hafsa Bint Bilal
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Neck Pain
Keywords: pain; proprioception; blood pressure; respiratory rate; cervical manipulation
MeSH Terms: conditions — Neck Pain; Pain | interventions — Manipulation, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cervical manipulation (Experimental): in the cervical manipulation, provide a high velocity, low-amplitude manipulation to each subject's cervical spine.
  Interventions: Other: cervical manipulation
- conventional therapy (Active Comparator): * 15 mins moist hot pack
  * Neck Isometric exercise
  * hold for 5-8 seconds and repeat 10 times
  * Cervical range of motion
  * 10 repetitions of movement in rotation within pain free range
  Interventions: Other: conventional therapy

INTERVENTIONS:
Other: cervical manipulation — provide a high velocity, low-amplitude manipulation to each subject's cervical spine.
  Arms: cervical manipulation
Other: conventional therapy — 15 mins moist hot pack Neck Isometric exercise hold for 5-8 seconds and repeat 10 times Cervical range of motion 10 repetitions of movement in rotation within pain free range
  Arms: conventional therapy

SUMMARY:
Mechanical neck pain is known as one of the most common disorders in musculoskeletal system. In elderly population, prevalence of neck pain ranges up to 38% while point prevalence and lifetime prevalence ranges from 6% to 22% and 14.2% to 71% respectively . Neck pain is defined by the international association for the study of pain as: "Pain perceived as arising from anywhere within the region bounded superiorly by superior nuchal line, inferior by transverse line through the tip of first thoracic spinous process, and laterally by sagittal plane tangential to the lateral border of neck" . There are variable causes of neck pain like trauma, infections, inflammatory conditions, musculoskeletal conditions, rheumatic diseases, and congenital diseases . There are varying degrees of disability and activity limitation caused by neck pain, like work productivity reduction and decrease quality of life . People who have a sedentary lifestyle, poor occupational postures, students with poor posture, people involved in occupation like computer programming, clerical job workers and desk job works are more likely to suffer from mechanical neck pain . Most common cause of mechanical neck pain is muscle tightness, Upper trapezius and levator scapulae are the most involved muscles

DETAILED DESCRIPTION:
Neck pain can over time negatively affect the central processing of any afferent input received because it can create a disturbance in the proprioceptive input to the Central Nervous System. Vuillerme stated that cervical muscle proprioceptors are stimulated by painful electrical stimuli. Therefore, joint proprioception can be affected in patients with mechanical neck pain .

The conservative management of mechanical neck pain includes many treatment options like electrotherapy which includes moist heat, Transcutaneous Electrical Nerve Stimulation therapy and different manual therapy options like cervical and thoracic mobilization and manipulation, Natural Apophyseal Glides and Sustained Natural Apophyseal Glides, Cyriax technique, manual pressure release, ischemic compression and proprioceptive neuromuscular facilitation. Postural reeducation and strength training of weak muscle group has beneficial effects. Joint mobilization and manipulation are widely used as a treatment for mechanical neck pain, as cervical mobilizations which are low velocity passive oscillatory movements are used by 90% of physiotherapist and chiropractors to treat people with neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-radiating neck pain of moderate intensity scoring 4-8 on the numeric pain rating scale (NPRS)
* Have a Neck Disability Index (NDI) score of 20% or greater (10 points or greater on a 0-to-50 scale)
* Patients who have cervical joint position error greater than 7.1 cm or 4.5 degrees

Exclusion Criteria:

* Patients with a positive history of trauma, fracture or surgery of the cervical spine .
* anatomical cervical spine abnormality
* presented with any neurological signs
* history of benign paroxysmal positional vertigo
* Neck pain with radiation to the arm and upper extremity .
* Diagnosed cases of torticollis, and scoliosis
* History of osteoporosis, Any cardiac disorder
* had participated in a neck exercise program in the past 6 months .

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
Joint position sense test | four weeks
  A target is placed on a wall 90cm away from the patient, at the patient's head height in sitting. The target is typically 40cm in diameter with concentric circles in 1cm increments. A laser pointer or similar targeting device is mounted onto a lightweight headband is then placed on the patient's head. The patient is then asked to focus on finding natural resting head position so that the laser pointer is in line with the center or "bullseye" of the target. With eyes closed, the patient will actively move their head in one plane of motion and attempt to return to the starting position as accurately as possible.
Digital sphygmomanometer | four weeks
  It is the most technologically advanced sphygmomanometer. It consists of an electronic sensor to measure the blood pressure and the readings are displayed on the digital monitor. To measure the blood pressure, the instrument measures the fluctuations of arteries
Respiratory rate measurement | four weeks
  To measure the respiratory rate of a person, ask the person to rest quietly for a moment. Start a timer for 60 seconds and count every time they breathe. Use the second hand on your watch or a timer on your phone to keep track of the person's breathing for exactly 1 minute. Once the minute starts, count every time you see their chest rise .
NPRS (Numeric Pain Rating Scale). | four weeks
  The Numeric Pain Rating Scale (NPRS) measures the subjective intensity of pain. The NPRS is an eleven-point scale from 0 to 10. "0" = no pain and "10" = the most intense pain imaginable while the NPRS exhibited moderate reliability
NDI (U) (Neck Disability Index) | four weeks
  The neck disability index is a ten-item self-reported questionnaire that assesses pain and associated disability, with a total max score of 50 points. An Urdu version of neck disability index will be used in this study. An intra-class correlation coefficient (ICC) revealed excellent test-retest reliability for all items (ICC = 0.86-0.98) and total scores (ICC = 0.99) of the NDI-U

CONTACTS AND LOCATIONS:
Overall Officials: maria Khalid, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah international hospital Sihala, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No